CLINICAL TRIAL: NCT04836260
Title: Preemptive Use of Convalescent Plasma for High-risk Patients With SARS-CoV-2 Infection: Phase III-IV Non-controlled Non-randomised Swiss Multicentric Trial
Brief Title: Preemptive Use of Convalescent Plasma for High-risk Patients With COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Ospedale Regionale di Lugano (Other); Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Diem-Lan Vu, MD, PhD, University Hospital, Geneva
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-02989
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Immuno-Deficiency; Old Age; Debility
Keywords: SARS-CoV-2; Convalescent plasma
MeSH Terms: conditions — COVID-19; Frailty | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: open-label non-controlled, non-randomised interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: SARS-CoV-2 convalescent plasma — Included patients will receive at least one unit of convalescent plasma with NTAB titer ≥1:160 at maximum 3-7 days after diagnosis by RT-PCR or symptom onset. A second unit of plasma from a different donor can be proposed 24h after the first unit if immunocompromised and/or the patient received less than 3-5ml/kg of plasma volume. Additional units can be exceptionnally infused, at the investigator discretion.

SUMMARY:
Convalescent plasma therapy has been recognized as safe and plasma transfusion is routinely used in clinical practice. A recent study showed that early administration of convalescent plasma can decrease the risk of complications in specific high-risk population.

The aim of the present study is to offer convalescent plasma therapy to immunocompromised patients and older adults in the early phase of a SARS-Cov-2 infection in order to accelerate viral clearance and prevent complication

DETAILED DESCRIPTION:
This is an open-label non-controlled, non-randomised interventional study. Study population consist in immunocompromised patients and older adults with or without co-morbidities.

Included patients will receive at least one unit of convalescent plasma with NTAB titer ≥1:160 or equivalent at maximum 3-7 days after diagnosis by RT-PCR or symptom onset or if having mild-moderate disease (WHO scale <4).

Patients will be followed-up up to 28 days to assess progression to WHO scale 4 disease, and 28-days mortality and viral load kinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Immunocompromised patients defined as

   1. Solid organ transplant ≤1 year before inclusion or treated for acute or chronic rejection episode or
   2. Allogeneic stem cell transplant recipients ≤2 years before inclusion or treated for acute GvHD ≥grade 2 or chronic moderate-severe GvHD or
   3. Active solid or haematological oncological disease with curative perspectives or
   4. HIV infection with CD4<350 or
   5. Hypogammaglobulinemia and other severe genetic immunological defect or
   6. Auto-immune disease with biological immunosuppressive treatment* or
   7. Other significant immunosuppressive condition such as IgG <6, treamtent with Rituximab or other biological lymphopenic treatment AND

      * Age ≥ 18 years old and
      * 2 distinct ABO group determination and
      * Positive RT-PCR for SARS-CoV-2 on a respiratory tract sample of ≤ 7 days and days post symptom onset (DPOS) ≤ 7 days at inclusion and/or
      * No oxygen requirement (WHO 8 ordinal scale < 4): asymptomatic, mild or moderate disease, or O2 saturation ≥ 90% at room temperature and
      * Compatible ABO donor with neutralizing antibodies (NTAB) ≥1 :160 or equivalent according to predefined antibody commercial assays cut-offs (see Study procedures)
      * RT-PCR on a respiratory tract sample with CT value<20 or ascending kinetics at the time of infusion (highly suggested but not necessary)
2. Older adults defined as Age ≥ 75 years old or ≥ 65 years old with at least one co-existing condition

   * Arterial hypertension under pharmacological treatment
   * Diabetes in treatment
   * Obesity (BMI ≥ 30 kg/m2)
   * Chronic obstructive pulmonary disease stade GOLD ≥2
   * Respiratory insufficiency due to any pneumopathy or neurologic disease.
   * Cardiovascular disease as defined by either known coronary heart disease, history of ischemic or hemorrhagic stroke or cardiac insufficiency (ejection fraction <40%)
   * Chronic kidney disease (GFR<60 ml/min) AND
   * 2 distinct ABO group determination and
   * Positive RT-PCR for SARS-CoV-2 on a respiratory tract sample of ≤ 3 days and days post symptom onset (DPOS) ≤ 3 days at inclusion or RT-PCR on a respiratory tract sample with CT value<20 or ascending kinetics at the time of perfusion and
   * No additional oxygen requirement compared to baseline (WHO 8 ordinal scale < 4): asymptomatic, mild or moderate disease and
   * Compatible ABO donor with neutralizing antibodies (NTAB) ≥1 :160 or equivalent according to predefined antibody commercial assays cut-offs (see Study procedures)

Exclusion criteria:

Seroconversion at the time of inclusion

* Palliative care
* No signed informed consent
* History of previous transfusion-related Grade 3 adverse event according to Swissmedic definitions
* Disseminated intravascular coagulopathy (depending on specialist evaluation)
* Uncontrolled acute hypervolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-08 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient that progress to WHO 8 ordinal scale ≥ 4 (oxygen requirement) | 7 days after plasma infusion
Proportion of patient that progress to WHO 8 ordinal scale ≥ 4 (oxygen requirement) | 14 days after plasma infusion
Proportion of death | 28 days after plasma infusion

SECONDARY OUTCOMES:
Proportion of patients with cleared nasopharyngeal viral load | 7 days after plasma infusion
  Cleared viral load is defined as CT value ≥30
Proportion of patients with cleared nasopharyngeal viral load | 14 days after plasma infusion
  Cleared viral load is defined as CT value ≥30

OTHER OUTCOMES:
Proportion of patients that progress to WHO 8 ordinal scale ≥ 4 (oxygen requirement) | 21 days after plasma infusion
Proportion of patients with cleared nasopharyngeal viral load | 21 days after plasma infusion
  Will be evaluated if CT< 30 at 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Kaiser, MD, Principal Investigator — University Hospital, Geneva; Enos Bernasconi, MD, Principal Investigator — Ospedale Regionale di Lugano; Véronique Erard, MD, Principal Investigator — HFR-Fribourg Hôpital Cantonal; Maja Weisser, MD, Principal Investigator — Klinik Infektiologie & Spitalhygiene
Locations (4):
- Switzerland (4):
  - Universitätsspital Basel, Basel
  - HFR-Fribourg Hôpital Cantonal, Fribourg
  - Geneva University Hospitals, Geneva
  - Ospedale Regionale di Lugano, Lugano

IPD SHARING:
Plan to Share IPD: Undecided